CLINICAL TRIAL: NCT03646630
Title: Ultrasound Guided Quadratus Lumborum Block Versus Caudal Block for Pain Relief in Children Undergoing Lower Abdominal Surgeries
Brief Title: Quadratus Lumborum Block Versus Caudal Block for Pediatric Postoperative Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University Hospital (Other)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, Doaa Lotfy, Assistant Lecturer of Anesthesiology, Fayoum University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: D141
Record Dates: First submitted 2018-08-01; First posted 2018-08-24 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Pain, Postoperative
Keywords: lower abdominal surgeries; quadratus lumborum block; caudal block
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quadratus Lumborum Block (QL) (Active Comparator): Patients will be placed in the lateral position,The high-frequency linear probe will be placed on the lateral abdomen, slightly cephalic to the iliac crest. Once the QL muscle will be observed, the probe will be tilted slightly to the caudal direction, to show the largest slice of the QL muscle, to confirm its posterior aspect. A 22-G block needle (Stimuplex D, Braun, Hongo, Bunkyo-ku, and Tokyo) will be inserted in-plane, ~1 cm ventral to the probe. The needle tip will be advanced until it penetrates the posterior fascia of the QL muscle. A small amount of saline will be injected to confirm the correct position of the tip, between the QL muscle and the erector spinae and latissimus dorsi muscles (Posterior or QL block type 2), then a bolus of 0.5 ml/Kg bupivacaine 0.25% will be injected.
  Interventions: Procedure: Quadratus Lumborum Block
- Caudal block (C) (Active Comparator): After induction of general anesthesia, a lateral position is obtained with the upper hip flexed 90⁰ and the lower one only 45⁰. A line is drawn to connect the posterior superior iliac spines bilaterally and used as one side of an equilateral triangle; then the location of the sacral hiatus should be approximated. By palpating the sacral cornua as 2 bony prominences, the sacral hiatus could be identified as a dimple in between. A 22 gauge needle is inserted at 45 degrees to the sacrum and redirected if the posterior surface of sacral bone is contacted. Children will receive caudal block with 1 ml/kg of bupivacaine 0.25%.
  Interventions: Procedure: Caudal Block

INTERVENTIONS:
Procedure: Quadratus Lumborum Block — Posterior or QL block type 2 , a bolus of 0.5 ml/Kg bupivacaine 0.25%
  Arms: Quadratus Lumborum Block (QL)
Procedure: Caudal Block — caudal block with 1 ml/kg of bupivacaine 0.25%.
  Arms: Caudal block (C)

SUMMARY:
The aim of this study is to compare between two regional analgesic techniques; caudal block and ultrasound guided quadratus lumborum block as regard degree of pain relief, accuracy of block, effect on hemodynamic stability and incidence of complications.

DETAILED DESCRIPTION:
Regional anesthesia and analgesia techniques are commonly used during pediatric surgical practice to facilitate pain control, decrease parenteral opioid requirements and improve the quality of post-operative pain control and patient-parent satisfaction. The most commonly used technique is caudal anesthesia, which is generally indicated for urologic surgery, inguinal hernia repair and lower extremity surgery. The quadratus lumborum (QL) block is a recently introduced abdominal truncal block, used for somatic and visceral analgesia of both the upper and lower abdomen. It was first described by Blanco in 2007 . Currently, the QL block is performed as one of the perioperative pain management procedures for all generations (pediatrics, pregnant, and adult) undergoing abdominal surgery . QL block allows the local anesthetics to spread between the posterior aspect of the quadratus lumborum muscle and the medial layer of the thoracolumbar fascia, which is close to the thoracic paravertebral space .

The ultrasound (US) has gained popularity among anesthesiologists performing regional anesthesia. Block success, and hence the efficacy would depend on the patient's anatomical variations and the anesthesiologist's skill level .

The use of ultrasound-guidance for peripheral nerve blocks (PNBs) offers many advantages. Direct visualization of the nervous and surrounding structures decreases the incidence of complications e.g. inadvertent intraneural or intravascular injection. Direct real-time observation of the local anesthetics spread ensures more accurate deposition .This leads to faster onset and longer duration of block, thus improves block quality. It also allows dose reduction of local anesthetics . It has been shown that when peripheral nerves are adequately imaged by ultrasound, the simultaneous use of the nerve stimulator offers no further advantages.

Following ethical committee approval of Anesthesia department, Fayoum University and obtaining informed consent from parents of each patient, fifty two patients will be randomized into 2 study groups. Each group contains 26 patients.

Methodology:

Preoperative Assessment:

All patients will be assessed clinically and investigated for exclusion of any of the above mentioned contraindications.

Operating Room Preparation & Equipment:

The ultrasound used will be Sonosite M Turbo (USA), the scanning probe will be the linear multi-frequency 13-6 MHz transducer (L25x13-6 MHz linear array). The needle used will be the stimuplex D needles manufactured by B Braun (Germany).

Perioperative Management:

All patients will be premedicated with IM midazolam 0.2 mg/kg and atropine 0.02 mg/kg. Perioperative monitoring will include continuous ECG, pulse oximetry, non-invasive arterial blood pressure, and temperature monitoring.

Inhalational induction of general anesthesia (GA) will be performed with a face mask using sevoflurane 8% and 50% oxygen in air, and then an intravenous (IV) cannula will be inserted. Fentanyl will be administered intravenously at 1 μg/kg, and a laryngeal mask airway (Intavent - Orthofix, Maidenhead, United Kingdom) will be used to secure the upper airway, with the patient kept spontaneously breathing. Anesthesia will be maintained with Isoflurane and 50% oxygen in air.

Surgery will be allowed to begin 10 minutes after block application. At the end of surgery, acetaminophen 15 mg/kg IV will be administered to all patients. Any complications occurring during the procedure will be recorded.

After completion of surgical procedure and emergence from anesthesia the patient will be referred to PACU. Quality of analgesia will be assessed using a FLACC scale at 30 minutes and at 1, 2, 4, 6, 12, and 24 hours postoperatively. Diclofenac sodium 1 mg/kg rectally will be given as rescue analgesia for patients in all study groups in PACU if FLACC scale > 4. Parents will be informed about the pain evaluation, and when patients had pain at home, parents will be instructed to give oral paracetamol 30 mg/kg. The anesthesiologist will record data received from the parents over the phone.

Statistical Analysis Sample size was calculated using the G* Power software version 3.1.7 analysis program (Heinirch Heine University, Dusseldorf, Germany) before the study. Depending on previous similar research with calculated effect size (d) 0.85, two tails (two sided), type 1 error 0.05 and increasing power of study to 90%, it was determined that each group should include at least 26 subject to obtain significant statistical value.

Collected data will be computerized and analyzed using statistical package for social science (SPSS) version 16. The results will be expressed as number and percentages for qualitative variables, mean, standard deviation and range for continuous data, median and inter-quartile range for quantitative discrete variables and scores.

To compare between groups, the chi-square will be used for qualitative variables, student t rest for comparing quantitative continuous variables between 2 groups, Mann Whitney U test to compare scores between 2 groups. Probability (P) value of less than 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Age 1-7 years
* American Society of Anesthesiologists physical status I-II
* Lower abdominal surgery

Exclusion Criteria:

* History of developmental delay or mental retardation
* Parent refusal
* History of allergic reactions to local anesthetics
* Rash or infection at the injection site
* Anatomical abnormality
* Bleeding disorders.
* History of cardiac, neurological, renal, hepatic diseases.

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2019-05-02 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
Time at which the first analgesia required | 24 hours after procedure
  in hours

SECONDARY OUTCOMES:
Pain assessment by the aid of FLACC score | 30 minutes after operation
  F:Face ,L:Legs, A:Activity, C:Cry, C:Consolability score
Pain assessment by the aid of FLACC score | 1 hour after operation
  F:Face ,L:Legs, A:Activity, C:Cry, C:Consolability score
Pain assessment by the aid of FLACC score | 2 hours after operation
  F:Face ,L:Legs, A:Activity, C:Cry, C:Consolability score
Pain assessment by the aid of FLACC score | 4 hours after operation
  F:Face ,L:Legs, A:Activity, C:Cry, C:Consolability score
Pain assessment by the aid of FLACC score | 6 hours after operation
  F:Face ,L:Legs, A:Activity, C:Cry, C:Consolability score
Pain assessment by the aid of FLACC score | 12 hours after operation
  F:Face ,L:Legs, A:Activity, C:Cry, C:Consolability score
Pain assessment by the aid of FLACC score | 24 hours after operation
  F:Face ,L:Legs, A:Activity, C:Cry, C:Consolability score
number of analgesic doses for each patient | 24 hours after operation
  by oral paracetamol 30 mg/kg given by parents
The general satisfaction score of parents | 24 hours after operation
  measured on a 5-point scale of 1.Extremely dissatisfied 2.Dissatisfied 3.Not satisfied, nor dissatisfied 4.Satisfied 5.Completely satisfied.
Preoperative heart rate | 5 minutes before operation
  in beat per minutes measured by electrocardiogram
Preoperative systolic blood pressure | 5 minutes before operation
  in mm mercury measured by non-invasive blood pressure measurement
Preoperative diastolic blood pressure | 5 minutes before operation
  in mm mercury measured by non-invasive blood pressure measurement
Intraoperative systolic blood pressure | every 15 minutes till end of operation
  in mm mercury measured by non-invasive blood pressure measurement
Intraoperative diastolic blood pressure | every 15 minutes till end of operation
  in mm mercury measured by non-invasive blood pressure measurement
Intraoperative heart rate | every 15 minutes till end of operation
  in beat per minutes measured by electrocardiogram
Incidence of hypotension | within one hour of the intervention
  drop of blood pressure more than 20 % of baseline blood pressure
Incidence of bradycardia | Within one hour of the intervention
  Heart rate below 50 beat per minute by electrocardiogram
Incidence of vascular puncture | Within one hour of the intervention
  as signs of local anesthetics toxicity
Incidence of convulsions | Within one hour of the intervention
  as signs of local anesthetics toxicity
Incidence of arrhythmias | Within one hour of the intervention
  as signs of local anesthetics toxicity
Incidence of paresthesia | Within one hour of the intervention
  as signs of local anesthetics toxicity
Incidence of hematoma formation | Within one hour of the intervention
  Recorded under ultrasound guidance
Incidence of injury to the underlying structures | Within one hour of the intervention
  Injury to the liver or a viscous

CONTACTS AND LOCATIONS:
Overall Officials: Kareem M Nawwar, MD, Study Director — Kasr ElAini Hospital, Faculty Of Medicine, Cairo Univerisity
Locations (1):
- Fayoum University hospital, El Fayoum Qesm, Faiyum Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kehlet H, Holte K. Effect of postoperative analgesia on surgical outcome. Br J Anaesth. 2001 Jul;87(1):62-72. doi: 10.1093/bja/87.1.62. No abstract available. PMID 11460814
- [Background] Willard FH, Vleeming A, Schuenke MD, Danneels L, Schleip R. The thoracolumbar fascia: anatomy, function and clinical considerations. J Anat. 2012 Dec;221(6):507-36. doi: 10.1111/j.1469-7580.2012.01511.x. Epub 2012 May 27. PMID 22630613
- [Background] Chakraborty A, Goswami J, Patro V. Ultrasound-guided continuous quadratus lumborum block for postoperative analgesia in a pediatric patient. A A Case Rep. 2015 Feb 1;4(3):34-6. doi: 10.1213/XAA.0000000000000090. PMID 25642956
- [Background] Liu SS, Ngeow J, John RS. Evidence basis for ultrasound-guided block characteristics: onset, quality, and duration. Reg Anesth Pain Med. 2010 Mar-Apr;35(2 Suppl):S26-35. doi: 10.1097/AAP.0b013e3181d266f0. PMID 20216022
- [Background] Griffin J, Nicholls B. Ultrasound in regional anaesthesia. Anaesthesia. 2010 Apr;65 Suppl 1:1-12. doi: 10.1111/j.1365-2044.2009.06200.x. PMID 20377542